CLINICAL TRIAL: NCT04669002
Title: Phase 2 Study to Evaluate the Safety & Efficacy of EP0057 in Combination With Olaparib in Advanced Ovarian Cancer Patients Who Have: Cohort 1 - Platinum Resistant Disease; Cohort 2 - Had at Least 1 Prior Line of Therapy Which Must Include at Least 1 Line of Platinum-based Chemotherapy Followed by PARP Inhibitor Maintenance
Brief Title: EP0057 in Combination With Olaparib in Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ellipses Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP0057-201
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer
Keywords: EP0057; Olaparib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 2A Cohort 1 (Experimental): Patients with advanced platinum resistant ovarian cancer who have received no more than 1 prior line of therapy which must be platinum-based chemotherapy
  Interventions: Drug: EP0057; Drug: Olaparib tablets
- Phase 2A Cohort 2 (Experimental): Patients with advanced ovarian cancer who have received at least 1 prior line of therapy which must include at least 1 line of platinum-based chemotherapy followed by a PARP inhibitor as maintenance treatment as their last treatment regimen
  Interventions: Drug: EP0057; Drug: Olaparib tablets

INTERVENTIONS:
Drug: EP0057 — EP0057 is an investigational nanoparticle-drug conjugate with a Camptothecin payload, that is administered intravenously
Drug: Olaparib tablets — Olaparib is a PARP inhibitor (poly [adenosine diphosphate-ribose] polymerase inhibitor)
  Other Names: Lynparza

SUMMARY:
EP0057-201 is a Phase 2A/B adaptive design study. Phase 2A will test EP0057 in combination with Olaparib and Phase 2B, the randomised part of the study, will test EP0057 in combination with Olaparib against SOC chemotherapy. When EP0057 is combined with Olaparib, it is envisaged that the combination should improve therapeutic responses in the recurrent ovarian cancer disease setting.

EP0057 is an investigational nanoparticle-drug conjugate administered intravenously. The rationale for developing EP0057 is to enable selective entry of EP0057 into tumour tissue and as a result create preferential accumulation of EP0057, and therefore of the payload Camptothecin, to translate into maximum tumour cell killing.

DETAILED DESCRIPTION:
EP0057-201 is an adaptive Phase 2A/B study in patients with advanced ovarian cancer.

Phase 2A

Phase 2A will be comprised of 2 single-arm treatment cohorts:

Cohort 1 will explore EP0057 in combination with Olaparib in patients with advanced platinum resistant ovarian cancer (see inclusion criteria for definition of platinum resistant) who have received no more than 1 prior line of therapy which must be platinum-based chemotherapy (n~=30)

Cohort 2 will explore EP0057 in combination with Olaparib in patients with advanced ovarian cancer who have received at least 1 prior line of therapy which must include at least 1 line of platinum-based chemotherapy followed by a PARP inhibitor as maintenance treatment as their last treatment regimen (n~=30)

It is anticipated that up to approximately 60 patients (approximately 30 patients per cohort) will be enrolled into Phase 2A. Both treatment cohorts will open in parallel and patients will be enrolled into each cohort concurrently.

At the end of Phase 2A, the Safety Review Committee will guide the decision to initiate 1 or both cohorts in Phase 2B, or terminate further recruitment into the study.

Phase 2B

Phase 2B will be comprised of 2 treatment cohorts, each randomised versus SOC. One or both cohorts may be opened concurrently to recruitment:

Cohort 1 will explore EP0057 in combination with Olaparib compared with SOC chemotherapy (TBC) in patients with advanced platinum resistant ovarian cancer who have received no more than 1 prior line of therapy which must be platinum-based chemotherapy (n=~132)

Cohort 2 will explore EP0057 in combination with Olaparib compared with SOC chemotherapy (TBC) in patients with advanced ovarian cancer who have received at least 1 prior line of therapy which must include at least 1 line of platinum-based chemotherapy followed by a PARP inhibitor as maintenance treatment as their last therapy (n=~192)

It is anticipated that ~324 patients will be enrolled into Phase 2B. Both treatment cohorts may open in parallel and patients may be enrolled into each cohort concurrently.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years of age at the time of Informed Consent
2. Ability to understand and provide written informed consent prior to undergoing any study procedures
3. Life expectancy of > 3 months, as estimated by the investigator
4. Histologically confirmed diagnosis (cytology alone excluded) with high-grade serous ovarian cancer or high-grade endometrioid ovarian cancer, including primary peritoneal or fallopian tube cancer
5. BRCA mutational status is known (germline and somatic). (For Patients in Phase 2A, status does not need to be known prior to enrolment)
6. HRD status is known. (For Patients in Phase 2A, status does not need to be known prior to enrolment)
7. At least 1 measurable lesion to assess response by RECIST v1.1 criteria
8. Archival tumour sample must be available. In the absence of an archival tumour biopsy, a tumour tissue biopsy will need to be collected prior to enrolment
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 at screening
10. Normal organ and bone marrow function:

    Haemoglobin ≥ 9.0 g/dL

    Absolute neutrophil count (ANC) ≥ 1.5 x 109

    Lymphocyte count ≥ 0.5 x 109

    Platelet count ≥ 100 x 109

    Total bilirubin ≤ 1.5 institutional upper limit normal (ULN)

    Serum albumin ≥ 2.5 g/dL

    AST and ALT ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN

    Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance > 50 mL/min (calculated using the Cockroft-Gault formula) for patients with creatinine levels above institutional normal

    Patients not receiving anti-coagulant medication must have an INR of ≤ 1.5 and an aPTT ≤ 1.5 x ULN
11. In the opinion of the Investigator, all other relevant medical conditions must be well-managed and stable for at least 28 days prior to first administration of study drug
12. Willing and able to participate in all required evaluations and procedures in this study protocol
13. Contraception: Each female subject of childbearing potential must agree to use a highly effective method of contraception (i.e., a method with less than 1% failure rate per year [e.g., sterilization, hormone implants, hormone injections, some intrauterine devices, vasectomized partner, or combined birth control pills]) from screening until 6 months after the last dose of EP0057 or Olaparib, whichever was taken last. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative serum or urine pregnancy test within 24 hours prior to EP0057 dosing on Day 1 of each Cycle (and must not be lactating). Each female subject will be considered to be of childbearing potential unless she has been surgically sterilised by hysterectomy or bilateral tubal ligation/salpingectomy or has been postmenopausal for at least 1 year.

    Cohort 1 patients (Phase 2A and 2B) must be/have:
14. Received no more than 1 prior line of therapy which must be platinum-based chemotherapy
15. Primary Platinum Resistant after completion of first line platinum-based chemotherapy

    Cohort 2 patients (Phase 2A and 2B) must have:
16. Received at least 1 prior line of treatment, 1 of which must be platinum-based chemotherapy
17. Received a PARP inhibitor in the maintenance setting as their most recent treatment following a confirmed response by RECIST1.1 (CR or PR) to the last regimen which must be a platinum-based chemotherapy, with maintenance of response by PARP inhibitor lasting ≥ 6 months, with subsequent confirmed disease progression as defined by RECIST v1.1 criteria

Exclusion Criteria:

1. Non-epithelial tumour of the ovary, the fallopian tube or the peritoneum
2. Ovarian tumours of low malignant potential or low grade
3. Prior treatment with a topoisomerase I inhibitor
4. Potent inhibitors or inducers of CYP3A4
5. Concurrent treatment with Coumadin (Warfarin)
6. History of stroke, transient ischemic attack, or myocardial infarction, within 6 months prior to C1D1
7. Brain and/or leptomeningeal metastases that are symptomatic or untreated or that require current therapy. Brain imaging must not be older than 12 weeks (at the start of screening). Results with abnormal/unexpected findings of brain MRI should be discussed with the Medical Monitor as part of the screening process
8. Systemic anti-cancer therapy for the disease under study within 3 weeks or 5 half-lives, whichever is longer, of the first dose of study drug
9. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 2 toxicities, which in the opinion of the Investigator should not exclude the patient
10. Patients considered by the Investigator to be at a higher baseline risk for new onset cystitis
11. Patients with a history, or features suggestive, of bone marrow dysplasia or myelodysplastic syndrome (MDS) or acute myeloid leukaemia (AML)
12. Confirmed QTcF > 470 msec on screening ECG or congenital long QT syndrome
13. Receiving an investigational anti-cancer treatment concurrently or within 3 weeks or 5 half-lives of either the parent drug or any active metabolite, whichever is longer, prior to the first dose of study drug
14. Any evidence of severe or uncontrolled systemic conditions (e.g., severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
15. Hypersensitivity to EP0057 or any of its excipients
16. Known history of Human Immunodeficiency Virus infection (HIV) (testing is not required), active infection with SARS-CoV-2, hepatitis B virus (HBV) or hepatitis C virus (HCV) per institutional protocol. Testing for HBV or HCV status is not necessary unless clinically indicated or the patient has a history of HBV or HCV infection. All patients should be tested for an active SARS-CoV-2 infection with an approved diagnostic test kit
17. Malignant disease other than that being treated in this study, with the following exceptions:

    Malignancies that were treated curatively and have not recurred within 2 years prior to study treatment

    Completely resected basal cell and squamous cell skin cancers

    Any malignancy considered to be indolent and that has never required therapy

    Completely resected carcinoma in situ of any type
18. Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results
19. Any major surgical procedure (in the investigator's judgement) within 2 weeks of the first dose of study drug
20. Pregnant, likely to become pregnant, or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of gestation)
21. Palliative radiotherapy (e.g., for pain or bleeding) within 6 weeks prior to randomisation or patients who have not completely recovered previous radiotherapy (Grade ≥ 2) from the effects of previous radiotherapy
22. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Note: Patients with indwelling catheters (e.g.,PleurX) are allowed
23. Hypersensitivity or intolerance (due to safety or other reasons) to PARP inhibitors

    Cohort 1 patients (Phase 2A and 2B) who:
24. Have primary platinum refractory disease defined as progression during first line treatment with 4-6 cycles of platinum based chemotherapy

    Cohort 2 patients (Phase 2A and 2B) who:
25. Progress within 6 months during PARP inhibitor maintenance treatment
26. Progress after completion of PARP inhibitor maintenance treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 18 months
  Overall Response Rate as measured using RECIST1.1
Number of patients with treatment emergent adverse events as assessed by NCI CTCAE version 5 | Approximately 18 months
Number of patients with related treatment emergent adverse events as assessed by NCI CTCAE version 5 | Approximately 18 months
Number of patients with serious adverse events | Approximately 18 months

CONTACTS AND LOCATIONS:
Locations (21):
- United States (11):
  - University of California Irvine, Irvine, California
  - Florida Cancer Specialists and Research Institute, Lady Lake, Florida
  - Augusta University, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - North Shore Hematology Oncology Associates PC DBA New York Cancer and Blood Specialists, East Setauket, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke Cancer Center, Durham, North Carolina
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Sarah Cannon, Nashville, Tennessee
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
- Hungary (4):
  - St. Margit Hospital, Budapest
  - National Institute of Oncology, Budapest
  - University of Debrecen Clinical Center, Debrecen
  - Petz Aladár County Teaching Hospital, Győr
- United Kingdom (6):
  - Royal Shrewsbury Hospital, Shrewsbury, Shropshire
  - Addenbrooke's Hospital, Cambridge
  - University College Hospital, London
  - Guy's Hospital, London
  - Hammersmith Hospital, London
  - Royal Stoke Hospital, Stoke-on-Trent